CLINICAL TRIAL: NCT02331953
Title: Predictors of Postoperative Delirium in Elder Patients After Spine Surgery: Regional Cerebral Oxygen Saturation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0606
Record Dates: First submitted 2014-12-29; First posted 2015-01-06 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Delirium in Elder Patients After Spine Surgery
Keywords: spine surgery; cerebral oximetry; postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- delirium group: the patients with delirium after spine surgery
- no delirium group: the patients without delirium after spine surgery

SUMMARY:
Postoperative delirium is an important problem in patients undergoing major surgery. The incidence of delirium was 12.5% in the patients over 70 years old undergoing spine surgery. A study shows that a low preoperative regional cerebral oxygen saturation (rSO2) is associated with postoperative delirium after on-pump cardiac surgery. This same perturbation likely also increases the risk for postoperative delirium after spine surgery, although there are little data that have evaluated this hypothesis. Therefore, this observational study was designed to explore the relationship between perioperative rSO2 and the delirium in elderly patients undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the study will be 60 or older undergoing elective major spine surgery (expected operative time is more than 2 hrs).
2. Patients who can do the mini-mental state examination (MMSE), Confusion Assessment Method for the ICU (CAM-ICU) and Intensive Care Delirium Screening Checklist (ICDSC).
3. Patients who understand the nature of the study and are willing to sign the consent form

Exclusion Criteria:

1. Emergency surgery
2. Patients diagnosed with neurocognitive disorders or psychiatric diseases, thus, cannot check MMSE or communicate with other people (e.g. Alzheimer's dementia, alcohol abuse)
3. Patients diagnosed with cerebrovascular disorders (e.g. stroke, atherosclerotic stenosis of carotid artery, TIA)
4. Patients who cannot be followed up until 2 days after surgery

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
the predictive power of periopertiver rSO2 regarding postoperative delirium | up to 2days postoperative
  The presence and severity of delirium were assessed with Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) once a day. (1 day preopertive, 2 days postoperative.) The investigators plan to evaluate whether periopertive rSO2 can predict postoperative delirium in elder patients after spine surgery and to assess the predictive power of periopertiver rSO2 regarding postoperative delirium. Perioperative rSO2 was observed during surgery (an expected average of 2~3 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Seoul, South Korea